CLINICAL TRIAL: NCT05392049
Title: Comparative Effects of Bowen's and Post Isometric Relaxation Techniques on Pain, Range of Motion and Function in Patients With Temporomandibular Joint Disorder
Brief Title: Effects of Bowen's Therapy and Post Isometric Relaxation Techniques in Patients of Temporomandibular Joint Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0106
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular disorder; Post isometric relaxation; Temporomandibular joint pain
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen's therapy (Experimental): Bowens therapy will be given to 12 patients of temporomandibular joint disorder .
  Interventions: Other: Bowen's therapy
- Post isometric relaxation (Experimental): post isometric relaxation technique will be given to12 patients of temporomandibular joint disorder.
  Interventions: Other: Post isometric relaxation

INTERVENTIONS:
Other: Bowen's therapy — Bowens technique will be apply on patients of TMJ for 2 repetitions in 1 set, 4 sets in each session for 4 weeks.
  Arms: Bowen's therapy
Other: Post isometric relaxation — post isometric relaxation technique and jaw exercises (strengthen the weakened muscles, stretch the shortened muscles) with dosage 5 times/session, 5 sec rest and 2times/week for 4 weeks will apply on patients.
  Arms: Post isometric relaxation

SUMMARY:
the aim of this study to compare effects of Bowen's therapy and post isometric relaxation techniques on pain, range of motions and function in patients with TMJ disorder.

DETAILED DESCRIPTION:
Temporomandibular joint disorder is a very common and serious problem of mouth and face pain related condition that mostly effect in quality of life and compromise the daily functional activities of a patient. It can be caused by any trauma, biomechanical, neuromuscular and psychologically related problems. Patient may come in acute and chronic phase. Patient condition mostly vary and worsen day by day, it thoughts that TMJD going interval throw out the life span of patient. Medicine, physical therapy interventions and surgical procedures are use in treatment of TMJ disorder. This study will conducted the comparative effects of Bowen's and post-isometric relaxation techniques on pain, ROM and functions in TMJ patients.

The study would be randomized clinical trial. Total 24 subjects will be assigned randomly into two groups by using lottery methods. Baseline treatment will be same (ultrasound, tapping) in both groups. Group A will be treated by Bowen's therapy and Group B will be treated by post-isometric relaxation technique for 30 min session (2 sessions/week and total 4 weeks). Numeric Pain Rating Scale, maximum mouth opening inter-incisal rural and jaw functional limitation scale-20 would be used as an outcome measurement tool for pain, range of motion and function respectively. Measurement will be taken at Baseline and at the end of the 4th week's treatment session. After assessing the normality data will be analyzed by using parametric / nonparametric test.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Participant aged 20-50.
* Pain on function.
* Restricted jaw movement.
* Clicking, popping sound.
* Tenderness in muscle of mastication.
* Joint tenderness.
* With a restricted mandibular range of motion 40mmor less measured interincisal.

Exclusion Criteria:

* Systematic arthropathy such as.
* Rheumatoid arthritis
* Fracture of jaw or TMJ.
* Malignant history of face and jaw.
* Prevent history of jaw or TMJ surgery.
* Subject has/ had dental/ orthodontic treatment within the past 14 days

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
NPRS for pain | 4th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Maximum Mouth opening (Inter- incisal Rural) for rang of motion | 4th week
  Maximum mouth opening is a vital and objective clinical parameter for assessment of stomatognathic region and it represents the range of vertical mandibular range of movement.The distance between the upper central incisor and lower incisor determined by flexible intra-oral ruler ,it is valid and reliable tool for measure TMJ distance.
Jaw Functional Limitation Scale for functional activity | 4th week
  Jaw functional limitation is a 20 items,3 level functional scale mastication, vertical jaw mobility, emotional and verbal expression. NO LIMITATION'' score have 0 and SEVER LIMITATION '' have 10 score

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Lahore Dental care clinic samnabad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moleirinho-Alves PMM, Cebola PMTC, Dos Santos PDG, Correia JP, Godinho C, Oliveira RANDS, Pezarat-Correia PLC. Effects of Therapeutic and Aerobic Exercise Programs on Pain, Neuromuscular Activation, and Bite Force in Patients with Temporomandibular Disorders. J Pers Med. 2021 Nov 10;11(11):1170. doi: 10.3390/jpm11111170. PMID 34834522
- [Background] Madariaga VI, Jasim H, Ghafouri B, Ernberg M. Myogenous temporomandibular disorders and salivary markers of oxidative stress-A cross-sectional study. J Oral Rehabil. 2021 Jan;48(1):1-9. doi: 10.1111/joor.13100. Epub 2020 Oct 5. PMID 32979853
- [Background] de Paiva Bertoli FM, Bruzamolin CD, de Almeida Kranz GO, Losso EM, Brancher JA, de Souza JF. Anxiety and malocclusion are associated with temporomandibular disorders in adolescents diagnosed by RDC/TMD. A cross-sectional study. J Oral Rehabil. 2018 Oct;45(10):747-755. doi: 10.1111/joor.12684. Epub 2018 Jul 20. PMID 29972708
- [Background] Osiewicz MA, Lobbezoo F, Loster BW, Loster JE, Manfredini D. Frequency of temporomandibular disorders diagnoses based on RDC/TMD in a Polish patient population. Cranio. 2018 Sep;36(5):304-310. doi: 10.1080/08869634.2017.1361052. Epub 2017 Aug 9. PMID 28792365
- [Background] Lee K, Lewis GN. Short term relief of multisite chronicpain with Bowen Therapy: A double-blind, randomized controlled trial. J Bodyw Mov Ther. 2020 Oct;24(4):271-279. doi: 10.1016/j.jbmt.2020.06.025. Epub 2020 Jul 30. PMID 33218522
- [Background] Tanhan A, Ozer AY, Polat MG. Efficacy of different combinations of physiotherapy techniques compared to exercise and patient education in temporomandibular disorders: A randomized controlled study. Cranio. 2023 Jul;41(4):389-401. doi: 10.1080/08869634.2021.1909454. Epub 2021 Apr 5. PMID 33818314
- [Background] Ram HK, Shah DN. Comparative evaluation of occlusal splint therapy and muscle energy technique in the management of temporomandibular disorders: A randomized controlled clinical trial. J Indian Prosthodont Soc. 2021 Oct-Dec;21(4):356-365. doi: 10.4103/jips.jips_332_21. PMID 34810363
- [Background] Volkan-Yazici M, Kolsuz ME, Kafa N, Yazici G, Evli C, Orhan K. Comparison of Kinesio Taping and manual therapy in the treatment of patients with bruxism using shear-wave elastography-A randomised clinical trial. Int J Clin Pract. 2021 Dec;75(12):e14902. doi: 10.1111/ijcp.14902. Epub 2021 Oct 8. PMID 34547165
- [Background] Asquini G, Pitance L, Michelotti A, Falla D. Effectiveness of manual therapy applied to craniomandibular structures in temporomandibular disorders: A systematic review. J Oral Rehabil. 2022 Apr;49(4):442-455. doi: 10.1111/joor.13299. Epub 2022 Jan 17. PMID 34931336
- [Derived] Javed S, Bashir MS, Mehmood A, Noor R, Ikram M, Hussain G. Comparative effects of post isometric relaxation technique and Bowen's therapy on pain, range of motion and function in patients with temporomandibular joint disorder. BMC Oral Health. 2024 Jun 12;24(1):679. doi: 10.1186/s12903-024-04440-1. PMID 38867195